CLINICAL TRIAL: NCT02800408
Title: Comparison of Beta-cryptoxanthin Bioavailability From Biofortified Maize in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: PepsiCo, Inc. (Industry); CIMMYT (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2015-1607
Record Dates: First submitted 2016-06-07; First posted 2016-06-15 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: β-cryptoxanthin Bioavailability From Biofortified Maize in Humans

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Whole grain high-BCX maize (Experimental): Whole grain, high-beta-cryptoxanthin (BCX; orange) maize will be incorporated into two muffins to be fed daily for 12 days. Complementary diet will be low in carotenoids.
  Interventions: Other: Whole grain high-BCX maize
- Refined grain high-BCX maize (Experimental): Refined (degermed) grain, high-beta-cryptoxanthin (BCX; orange) maize will be incorporated into two muffins to be fed daily for 12 days. Complementary diet will be low in carotenoids.
  Interventions: Other: Refined grain high-BCX maize
- Whole grain white maize (Placebo Comparator): Whole grain, white maize (low in beta-cryptoxanthin) will be incorporated into two muffins to be fed daily for 12 days. Complementary diet will be low in carotenoids.
  Interventions: Other: Whole grain white maize

INTERVENTIONS:
Other: Whole grain high-BCX maize — The whole grain orange maize will be milled and prepared into muffins to be consumed daily. Muffins will contain a target of 500 µg beta-cryptoxanthin per day.
  Other Names: Whole grain high-beta-cryptoxanthin maize; Whole grain orange maize
  Arms: Whole grain high-BCX maize
Other: Refined grain high-BCX maize — The refined grain orange maize will be degermed, milled, and prepared into muffins to be consumed daily. Muffins will contain a target of 500 µg beta-cryptoxanthin per day.
  Other Names: Refined grain high-beta-cryptoxanthin maize; Refined grain orange maize
  Arms: Refined grain high-BCX maize
Other: Whole grain white maize — The whole grain white maize will be milled and prepared into muffins to be consumed daily. Muffins will contain minimal beta-cryptoxanthin, matched for dry maize weight.
  Other Names: Whole grain low-beta-cryptoxanthin maize
  Arms: Whole grain white maize

SUMMARY:
The purpose of this study is to determine how well the body absorbs the carotenoid beta-cryptoxanthin (BCX) from a type of corn that has been naturally bred (not genetically engineered) to contain higher amounts of BCX than traditional breeds of corn. Because this new type of corn contains higher amounts of BCX, it appears more orange in color than traditional types of corn. Understanding how well the body can absorb the BCX from the corn may help companies develop food products that may have improved nutritional quality.

DETAILED DESCRIPTION:
Randomized, blinded, 3 x 3 crossover intervention. Each treatment will last 12 d, followed by a 7-d wash-out period. After the washout, subjects will go back to their regular diet for two weeks before beginning the next cycle. Subjects will report to the research kitchen in the Nutritional Sciences building for their breakfast. Maize will be incorporated into two muffins. Other food choices will be yogurt and other low-fiber foods. Blood samples will be taken at baseline and days 3, 6, 9, 12, 15, and 19. Natural abundance measurements of 13-carbone to 12-carbon will be taken at baseline, day 12 and day 19. Retinol isotope dilution testing will be done at the end of the study to determine total body stores of vitamin A in the subjects. This will include the day 19 blood sample of intervention phase 3 and a final blood sample 14 days after the isotope dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 28 y, BMI 19 - 26 kg/m2, non-smoking, not pregnant or trying to become pregnant, and not lactating.

Exclusion Criteria:

* Smoker
* BMI < 19 kg/m^2 or BMI > 26 kg/m^2
* Women: pregnant or trying to become pregnant, breast-feeding
* Weight loss greater than or equal to 10 pounds (4.5 kilograms) during the 3 months prior to recruitment
* Actively trying to lose weight
* Fat malabsorptive disorders
* Inability to refrain from drinking alcohol when requested
* Amenorrhea
* Acute or chronic illness, including hepatitis
* Current or previous history of anorexia or bulimia
* History of iron deficiency anemia
* Inability to pick up food from research facility and eat meals on site when requested
* Planned vacation of >1 week duration during the study
* Known scheduling conflict with the blood draws
* Major food allergies/intolerance to ingredients used in the meals
* Unwillingness to discontinue personal nutritional supplements/vitamins when asked to
* Concurrent participation in other studies
* Social circumstances that would make it difficult to consume a study food
* Family member already enrolled in the study

Ages: 20 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2017-10-23 (Actual)

PRIMARY OUTCOMES:
Serum beta-cryptoxanthin concentration area under the curve ((µmol/L)*t) | 19 days with blood samples drawn on days 0, 3, 6, 9, 12, 15, 19 of treatment phase
  Serum beta-cryptoxanthin concentration area under the curve calculated from samples on days 0, 3, 6, 9, 12, 15, 19 of treatment phase

SECONDARY OUTCOMES:
Serum retinol carbon-13 natural abundance (δ 13C‰) | 19 days and will be measured on days 0, 12, and 19
  Change in serum retinol carbon-13 natural abundance will be assessed from beginning to after each treatment period. This will be done on baseline, day 12 and day 19 blood samples.
Vitamin A total body stores (µmol vitamin A) by retinol isotope dilution | 14 days and will include the final blood of phase three and another sample 14 days later
  After a blood draw, a carbon-13 labeled vitamin A oral dose will be given to subjects after all treatments. After 14 days, another blood draw will be taken to determine dilution of the stable isotope dose. This will used the final blood sample of intervention phase 3 and a final blood draw 14 days later.
Vitamin A estimated total liver reserves (µmol vitamin A/g liver) by retinol isotope dilution | 14 days and will include the final blood of phase three and another sample 14 days later
  After a blood draw, a carbon-13 labeled vitamin A oral dose will be given to subjects after all treatments. After 14 days, another blood draw will be taken to determine dilution of the stable isotope dose. This will used the final blood sample of intervention phase 3 and a final blood draw 14 days later.
Serum zeaxanthin, lutein, and beta-carotene concentration area under the curves ((µmol/L)*t) | 19 days with blood samples drawn on days 0, 3, 6, 9, 12, 15, 19 of treatment phase
  Serum carotenoid concentration area under the curves calculated from samples on days 0, 3, 6, 9, 12, 15, 19 of treatment phase

CONTACTS AND LOCATIONS:
Overall Officials: Sherry A Tanumihardjo, Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison Nutritional Sciences, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arscott SA, Simon PW, Tanumihardjo SA. Anthocyanins in purple-orange carrots (Daucus carota L.) do not influence the bioavailability of beta-carotene in young women. J Agric Food Chem. 2010 Mar 10;58(5):2877-81. doi: 10.1021/jf9041326. PMID 20131807
- [Background] Horvitz MA, Simon PW, Tanumihardjo SA. Lycopene and beta-carotene are bioavailable from lycopene 'red' carrots in humans. Eur J Clin Nutr. 2004 May;58(5):803-11. doi: 10.1038/sj.ejcn.1601880. PMID 15116084
- [Background] Molldrem KL, Li J, Simon PW, Tanumihardjo SA. Lutein and beta-carotene from lutein-containing yellow carrots are bioavailable in humans. Am J Clin Nutr. 2004 Jul;80(1):131-6. doi: 10.1093/ajcn/80.1.131. PMID 15213039
- [Background] Tanumihardjo SA, Horvitz MA, Dosti MP, Simon PW. Serum alpha- and beta-carotene concentrations qualitatively respond to sustained carrot feeding. Exp Biol Med (Maywood). 2009 Nov;234(11):1280-6. doi: 10.3181/0903-RM-106. Epub 2009 Aug 5. PMID 19657072
- [Background] Osth M, Ost A, Kjolhede P, Stralfors P. The concentration of beta-carotene in human adipocytes, but not the whole-body adipocyte stores, is reduced in obesity. PLoS One. 2014 Jan 8;9(1):e85610. doi: 10.1371/journal.pone.0085610. eCollection 2014. PMID 24416432
- [Result] Titcomb TJ, Sheftel J, Sowa M, Gannon BM, Davis CR, Palacios-Rojas N, Tanumihardjo SA. beta-Cryptoxanthin and zeaxanthin are highly bioavailable from whole-grain and refined biofortified orange maize in humans with optimal vitamin A status: a randomized, crossover, placebo-controlled trial. Am J Clin Nutr. 2018 Oct 1;108(4):793-802. doi: 10.1093/ajcn/nqy134. PMID 30321275